CLINICAL TRIAL: NCT05414214
Title: Thyromental Height Test Versus Sternomental Displacement Test for Prediction of Difficult Airway in Elderly Surgical Patients.
Brief Title: Thyromental Height Test Versus Sternomental Displacement in Elderly
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, assisstant professor, Cairo University
Other Study IDs: 45MS-2021
Record Dates: First submitted 2022-06-08; First posted 2022-06-10 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Difficult Airway
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly: Elderly patients who are scheduled for elective surgeries under general anesthesia with endotracheal intubation accomplished using conventional laryngoscopy will be included.
  Interventions: Procedure: Thyromental Height Test; Procedure: Sternomental displacement; Procedure: General anesthesia

INTERVENTIONS:
Procedure: Thyromental Height Test — Thyromental Height Test (TMHT) : will be measured while a patient is lying supine with the head and neck are maintained in a neutral position using a pillow under the head. By using a digital depth gauge, the TMH is the vertical distance measured between the anterior border of the thyroid cartilage directly on the thyroid notch and the anterior border of the mentum.
Procedure: Sternomental displacement — Sternomental displacement (SMDD): While the patient is sitting with the head in a neutral position, SMD-neutral will be measured using a tape as the distance between upper borders of the manubrium sterni and the mentum. The SMD-extension will then be measured in the same way with the head extended on the neck. The difference between SMD-extension and SMD-neutral will then be calculated as SMDD.
Procedure: General anesthesia — patients will be pre-oxygenated with 100% oxygen for 3 minutes, anesthesia will be then induced intravenously using fentanyl 2 μg/kg, propofol 1 -1.5 mg/kg, and succinylcholine 1 mg/kg lean body weight. Mask ventilation will be maintained till complete muscle relaxation guided by a peripheral nerve stimulator. Using Macintosh laryngoscopy, an anesthetist who has at least three years experience and who will be blinded to the preoperative tests' results, determined the best laryngeal view by using Cormack-Lehane (CL) grading system from I-IV. External neck manipulation will be used when needed to obtain the best laryngoscopic view. Endotracheal intubation will then be accomplished. The number and duration of intubation attempts will be recorded.

SUMMARY:
The study is designed to evaluate the validity of the SMDD as a predictor of difficult airway in elderly and to compare its validity with that of the TMHT.

DETAILED DESCRIPTION:
The airway assessment for difficulty before anesthesia in the elderly is crucial as the delay in the endotracheal intubation in this age group can lead to fatal consequences due to limited organ reserve and comorbidities. Previous studies revealed that elderly patients are predisposed to an increased incidence of difficult airway due to the age-related anatomic changes of the head and neck. These changes include, but not limited to, teeth loss, narrow dental arch, reduced oral soft tissue flexibility, TMJ dysfunction, degenerative change of ligament and tendons of the intervertebral discs causing compression of the intervertebral discs, cervical lordosis and spondylosis, limited head and upper neck extension, and fixed cervical spine flexion deformity.

Sternomental displacement (SMDD) is a relatively new objective airway measure that represents the difference between Sternomental distance that is measured while the head is extended on the neck (SMD-extension) and the Sternomental distance that is measured while the head is in a neutral position (SMD-neutral). The SMDD is a surrogate indicator of neck mobility. Both TMHT and SMDD were proved to be a good objective predictor for difficult laryngoscopy (DL) in adult surgical patients.

The TMHT was proved to have good predictive ability for difficult airway in elderly patients, but to the best of our knowledge, the SMDD was not previously evaluated in elderly. This study was designed to evaluate the validity of the SMDD as a predictor of difficult airway in elderly and to compare its validity with that of the TMHT. Our primary endpoint is the AUROC curve (area under receiver operating characteristic curve), sensitivity, specificity of the SMDD as a predictor of difficult laryngoscopy in elderly surgical patients. The secondary endpoint is to compare the validity of SMDD for predicting difficult airway with that of the TMHT and (Modified Mallampati test) MMT.

ELIGIBILITY:
Inclusion Criteria:

1. elderly patients aged ≥ 65 years both male & female .
2. ASA physical status I, II, and III .
3. patients scheduled for elective surgeries under general anesthesia .

Exclusion Criteria:

1. Patients undergoing emergency procedure
2. patients requiring elective awake fiberoptic.
3. patients having neuromuscular disorders or craniofacial abnormalities
4. patients with cervical spine surgeries, neck scars, obvious limited neck extension.
5. morbid obesity (MBI ˃40 kg/m2)

Ages: 65 Years to 90 Years | Sex: All
Age Groups: Older Adult
Study Population: In our study, 150 elderly patients who are scheduled for elective surgeries under general anesthesia with endotracheal intubation accomplished using conventional laryngoscopy will be included.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
sensitivity, specificity of the sternomental displacement as a predictor of difficult laryngoscopy in elderly surgical patients. | 10 minutes

SECONDARY OUTCOMES:
Thyromental Height Test (TMHT) | 10 minutes
  Thyromental Height Test (TMHT): will be measured while a patient is lying supine with the head and neck are maintained in a neutral position using a pillow under the head. By using a digital depth gauge, the TMH is the vertical distance measured between the anterior border of the thyroid cartilage directly on the thyroid notch and the anterior border of the mentum.
Sternomental displacement (SMDD) | 10 minutes
  Sternomental displacement (SMDD): While the patient is sitting with the head in a neutral position, SMD-neutral will be measured using a tape as the distance between upper borders of the manubrium sterni and the mentum. The SMD-extension will then be measured in the same way with the head extended on the neck. The difference between SMD-extension and SMD-
Modified Mallampati test (MMT) | 10 minutes
  Modified Mallampati test (MMT): the patient will be seated in a neutral position, the mouth is maximally opened, tongue protruded, and no phonation. According to the apparent oropharyngeal structures, the proper classification will be recorded.
Cormack-Lehane (CL) grading system | 10 minutes
  Cormack-Lehane (CL) grading system from I-IV. (Grade I: full view of the glottis; grade II: glottis partly exposed, anterior commissure not seen; grade III: only epiglottis seen; grade IV: epiglottis not seen). Grade I &II will be categorized as easy laryngoscopy and grade III and IV as difficult laryngoscopy.
The number and duration of intubation attempts | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Ahmed, MD, Principal Investigator — Cairo University
Locations (1):
- Faculty of medicine-Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson KN, Botros DB, Groban L, Bryan YF. Anatomic and physiopathologic changes affecting the airway of the elderly patient: implications for geriatric-focused airway management. Clin Interv Aging. 2015 Dec 4;10:1925-34. doi: 10.2147/CIA.S93796. eCollection 2015. PMID 26673904
- [Background] Etezadi F, Ahangari A, Shokri H, Najafi A, Khajavi MR, Daghigh M, Moharari RS. Thyromental height: a new clinical test for prediction of difficult laryngoscopy. Anesth Analg. 2013 Dec;117(6):1347-51. doi: 10.1213/ANE.0b013e3182a8c734. PMID 24257384
- [Background] Prakash S, Mullick P, Bhandari S, Kumar A, Gogia AR, Singh R. Sternomental distance and sternomental displacement as predictors of difficult laryngoscopy and intubation in adult patients. Saudi J Anaesth. 2017 Jul-Sep;11(3):273-278. doi: 10.4103/1658-354X.206798. PMID 28757825